CLINICAL TRIAL: NCT03002051
Title: EUS-guided Transenteric Drainage With a Novel Lumen-apposing Metal Stent for the Management of Pancreato-biliary Diseases: a Multi-national, Multicenter Prospective Study
Brief Title: EUS-guided Transenteric Drainage With a Novel Lumen-apposing Metal Stent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: SoonChunHyang University School of Medicine (Unknown)
Responsible Party: Principal Investigator, Anthony Teoh, Associate Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPAXUS version 3.0
Record Dates: First submitted 2016-12-16; First posted 2016-12-23 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Pancreatic Pseudocyst; Pancreatic Necrosis; Biliary Obstruction; Acute Cholecystitis
MeSH Terms: conditions — Pancreatic Pseudocyst; Pancreatitis, Acute Necrotizing; Cholecystitis, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EUS guided drainage (Experimental): Patients suffering from the conditions in focus would receive EUS guided drainage with the lumen apposing stent
  Interventions: Device: EUS-guided drainage

INTERVENTIONS:
Device: EUS-guided drainage — * Ultrasonographic evaluation of the lesion by linear echoendoscope and positioning for transenteric puncture in shortest distance between enteric wall and the target lumen for drainage.
  * EUS-guided transenteric puncture by using a 19-gauge needle followed by placement of a 0.035 or 0.025-inch guidewire into the target lumen.
  * After the needle is removed in remaining the guidewire, the tract is dilated over the guidewire by using bougie dilator or needle type cystotome (Endoflex, Voerde, Germany). And then, the tract may be more dilated by using balloon catheter (4-mm).
  * After dilation of the tract, stent delivery system is inserted over the guidewire into the target lumen.
  * After complete deployment of the distal flange under EUS and fluoroscopic guidance into the target lumen, proximal retraction of the delivery system until the blue mark on the handle of the introducer is seen. And then, the proximal flange is deployed slowly under endoscopic guidance.

SUMMARY:
To evaluate clinical efficacy and safety of a novel lumen-apposing FCSEMS for EUS-guided transenteric drainage of PFC or of biliary tree including GB

DETAILED DESCRIPTION:
Patients with the following conditions would be recruited for drainage under EUS guidance with the new lumen apposing FCSEMS

* Symptomatic or infected pancreatic pseudocyst or walled-off necrosis (WON) (SPAXUS 16 or 10 mm)
* Acute cholecystitis by inoperable malignant diseases (SPAXUS 10 mm)
* Acute cholecystitis by benign conditions with high-risk for operation (SPAXUS 10 mm)
* Long-term cholecystostomy at high-risk for operation (SPAXUS 10 mm)
* Symptomatic malignant obstruction of the distal CBD with unsuccessful transpapillary approach (the diameter of the CBD > 10 mm) (SPAXUS 8 or 10 mm)

Outcome paramaters include technical and clinical success, adverse events.

ELIGIBILITY:
Inclusion Criteria:

Patient must meet all of the following inclusion criteria to be eligible for enrollment into the study.

* Pancreatobiliary diseases that are eligible for EUS-guided transenteric drainage
* The patient who aged from 20 to 80 years. Legally acceptable representative must be capable of giving written informed consent prior to participation in this study
* Target lesion that is accessible through the transenteric approach
* The woman of child-bearing age must be negative from the pregnancy test in order to participate in this study
* The patient who is willing and able to comply with the scheduled visits, treatment plan, laboratory tests, and other study procedures
* The patients should not have any unacceptable conditions (e.g., physiological, familyism, social, geographical) for medical follow-up and adaptation of the study.

Exclusion Criteria:

Patient presenting with any of the following will not be included in the study.

* Inaccessible to EUS-guided approach
* Bleeding tendency: International normalized ratio (INR) of prothrombin time < 1.5 or platelet conunt < 60,000/mm3
* Patients with Disseminated Intravascular Coagulation syndrome(DIC)
* Patients who have been taking medicines that can cause hemorrhage (e.g., Aspirin, Wafarin etc.)
* Patients with other serious disease or medical condition
* Patients with past medical history of significant neurologic or Psychiatric disorders such as dementia or seizure
* Unstable heart disease despite of treatment, recent myocardial infarction within 6 month (Even though MI was diagnosed within 6 months, if it becomes stable presently, the patient can be possible to participate).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Clinical success for pancreatic fluid collections | 8 hrs
  ① Clinical success of pancreatic fluid collections
  * Peudocyst: resolution more than 50% in the initial size of cyst.
  * Walled-off necrosis: resolution of PFC without the need for additional interventions after endoscopic interventions.
Clinical success for acute cholecystitis | 8hrs
  - Afebrile for 8 hours, tolerating diet, absence of abdominal sign, or 20% decrease in white cell count.
Clinical success for obstructive jaundice | 2 weeks
  - A decrease in total bilirubin to < 50 % of the pre-stenting value within 2 weeks.

SECONDARY OUTCOMES:
Techincal success | 1 day
  - Satisfactory access, placement of stent and drainage.
Adverse events | 30 day
  * Bleeding: any hemorrhagic event during or after the procedure that required endotherapy, radiological interventions, blood product transfusion, or inpatient observation.
    * Perforation: perforation of the GI tract or cystic wall on imaging studies with peritonitis signs.
      * Pneumoperitoneum or pneumoretroperitoneum: intraperitoneal or retroperitoneal air on imaging study.
        * Stent migration: dislocation of the stent into the lumen or the GI tract on imaging study

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Teoh, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teoh AYB, Kongkam P, Bapaye A, Ratanachu T, Reknimitr R, Lakthakia S, Chan SM, Gadhikar HP, Korrapati SK, Lee YN, Medarapalem J, Ridtitid W, Moon JH. Use of a novel lumen apposing metallic stent for drainage of the bile duct and gallbladder: Long term outcomes of a prospective international trial. Dig Endosc. 2021 Nov;33(7):1139-1145. doi: 10.1111/den.13911. Epub 2021 Jan 11. PMID 33284467